CLINICAL TRIAL: NCT06726564
Title: A Phase 1 Single Arm, Dose Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of MT027 in Patients with Pleural Malignant Tumors
Brief Title: A Study of MT027 in Patients with Pleural Malignant Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Suzhou Maximum Bio-tech Co., Ltd. (Industry)
Collaborators: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MT027-MPE-001
Record Dates: First submitted 2024-06-11; First posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Advanced Malignant Solid Tumor; Malignant Pleural Effusion; Pleura Carcinoma; Pleural Mesothelioma; Pleural Malignant Mesothelioma; Pleural Metastases
Keywords: advanced malignant solid tumors; metastatic or primary malignant tumors in the pleural cavity; malignant pleural effusion
MeSH Terms: conditions — Pleural Effusion, Malignant; Mesothelioma, Malignant; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MT027 (Experimental)
  Interventions: Drug: MT027 cells suspension

INTERVENTIONS:
Drug: MT027 cells suspension — MT027: CRISPR/Cas9 edited B7H3-specific allogeneic CAR-T cells

SUMMARY:
This is a phase I open label, single-arm, dose-escalation study to evaluate the feasibility, safety, tolerability, PK/PD, and to determine RP2D of MT027 via an locoregional delivery in subjects with pleural malignant tumors, who have previously received standard of care therapy..

Subjects meeting the study entry criteria including having tumor antigen B7H3 overexpression via immunohistochemistry (IHC ) will be enrolled and assigned to cohorts sequentially to receive study treatments, assessments, as well as post-treatment safety follow-ups in the study.

DETAILED DESCRIPTION:
MT027 will be given intrapleural injection via pleural cavity puncture on Day 1 of the first 28-day cycle, followed by a 28-day DLT observation period. After the first cycle, if the subject does not experience any unacceptable toxicities and disease progress, additional treatment may be continued every three weeks thereafter. The second study drug injection of Cycle 2 will occur on one to two days after Day 28, and the subsequent study drug administrations will be on first or second day of each successive 21 day-cycle.

After receiving the first ICV administration of the study drug, the subject will be observed in the hospital with accessibility to bedside monitors and emergency care for a minimum of seven consecutive days, and discharged after the safety assessments are performed without safety concerns at the discretion of the PI. The subject will be further assessed for safety evaluation on Day14 and Day 28, prior to the initiation of the second injection . A shortened observation period may begin with the second injection at the discretion of the principal investigator (PI).

Subjects on-study will receive treatment until intolerable toxicity based on PI's clinical assessment , disease progression, voluntary withdrawal or death. Dose reduction of MT027 may be considered for optimal safety management of the subject, upon the discussion with the Sponsor Medical Monitor. Study drug may be temperately interrupted to allow safety management at the subject level and will resume the study treatment dose after patient's adverse events are recovered to the grade I level, per PI's discretion. Study drug treatment should be discontinued in the following circumstances: The Investigator considers that the subject will no longer benefit from the treatment; the subject develops intolerable toxicity or disease progression ; the subject withdraws the informed consent; or the subject is lost to follow-up.

Subjects who complete the study or withdraw from the study for any reason should be followed at the end of treatment/early termination (EOT/ET) within 30 days from the last study drug infusion or becoming aware of the study discontinuation. A telephone follow-up every 12 weeks post EOT/ET for a maximum of 15 years after the 1st dose will be performed, as deemed clinically necessary.

Dose escalation will follow a standard 3+3 design. Three dose levels will be explored. Dose escalation will depend on the proportion and intensity of observed toxicities. The number of CAR-T cells in a given cohort could be revised upon the data review of upcoming safety and PK/PD data during the study. The different dose level(s) could be implemented during the escalation phase, if clinically deemed necessary.

ELIGIBILITY:
Inclusion Criteria:

1. voluntarily participate in the study and sign informed consent;
2. age over 18 years old (including the cut-off value), regardless of gender;
3. advanced malignant solid tumor pathologically and/or histologically diagnosed with malignant pleural effusion requiring drainage confirmed by histopathology or cytopathology (metastatic or primary);
4. the original pleural cavity malignant tumor after standard treatment failure, or top treatment;
5. signed informed consent not line within a month before the chest cavity medicine injection, but does not exclude the diagnostic puncture;
6. The subjects voluntarily provided sufficient tumor cells in the pathological section of the primary lesion and/or pleural effusion for B7-H3 expression detection, and the tumor cells in the pathological section of the primary lesion or malignant pleural effusion were positive for B7-H3 expression;
7. Eastern Cooperative Oncology Group (ECOG) performance status (PS) score 0-2;
8. within 7 days before treatment laboratory meet the following criteria:

Routine blood (14 days) :

1. Absolute neutrophil count (ANC) ≥1.5×109 /L;
2. platelet count (PLT) or 80 x 109 / L;
3. hemoglobin (HGB) or 80 g/L (allowing blood transfusion and use erythropoiesis agent). The presence of active bleeding or other ongoing conditions that result in increased red-cell destruction or impaired production may require repeated transfusions or red-cell therapy, and patients had to discuss their eligibility with the sponsor on an individual basis before enrollment.) ;

Liver:

1. total bilirubin (TIBC) or less 2 times the upper limit of the normal range (ULN);
2. no liver metastasis, AST and ALT 3 x ULN or less; ALT and AST≤5 times ULN in the presence of liver metastasis;

Kidney:

1. Serum creatinine (Cr) ≤ 2 times ULN; Or creatinine clearance (CrCL) ≥ 50 mL/min (estimated by Cockcroft-Gault formula);

   Blood coagulation function:
2. international standardization ratio (INR) or prothrombin time (PT) 1.3 x ULN or less;
3. Partial activated thromboplastin time (APTT) ≤ 1.5 times ULN; 9) toxicity from previous systemic therapy returned to grade 1 or less or to baseline before the first dose (except alopecia); 10) Fertile men and women of childbearing age must agree to use reliable contraception from the time they provide informed consent until 180 days after the last dose of MT027 cell injection; Women of childbearing age included those who were premenopausal and those within 2 years of menopause.

Exclusion Criteria:

1. known allergy to the study drug or its excipients;
2. patients with pleural puncture contraindications or won't benefit from intrathoracic medication;
3. any antineoplastic drugs other than systemic antineoplastic therapy that the subject has been taking stably and any treatment that may have an effect on the control of pleural effusion (other than diagnostic puncture or thoracentesis for investigational treatment);
4. in the first test within 2 weeks before treatment received radiotherapy.
5. major surgery is performed within 4 weeks before the first trial treatment and the patient has not fully recovered;
6. are receiving systemic steroid therapy or any other form of immunosuppressive therapy within 1 week before the first trial treatment.
7. participated in other drug clinical trials within 4 weeks before screening;
8. always had targeted B7 - H3 CAR - T cells treatment;
9. patients with active systemic or pulmonary infection, coagulopathy and other major diseases;
10. with severe heart, lung, liver and renal insufficiency; Cardiac function: grade 3 or above according to the New York Heart Association (NYHA) criteria; Liver function: Child - Puge classification standard for grade C or above; Renal function: chronic kidney disease (CKD) stage 4 or above; Renal insufficiency stage Ⅲ or above; Pulmonary function: severe symptoms of respiratory failure involving other organs;
11. patients with severe autoimmune diseases;
12. recipients of previous allogeneic tissue/solid organ transplantation;
13. who received a live vaccine within 2 weeks before the first cell therapy or were scheduled to receive a live vaccine during the study;
14. active HBV infection; Or hepatitis C virus infection (defined as positive for HCV antibody, allowed if HCV-RNA was below the lower limit of detection); Or human immunodeficiency virus infection (defined as HIV antibody positive); Or positive treponema pallidum antibody;
15. subjects had severe neurocognitive impairment as judged by the investigator;
16. pregnant or lactating women;
17. There were any clinical or laboratory abnormalities or other reasons considered by the investigator to preclude participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
adverse events (AE) and serious adverse events (SAE) | through study completion, an average of 1 year
Dose Limiting Toxicity (DLT) | 28 days
GvHD | through study completion, an average of 1 year
CRS | through study completion, an average of 1 year
Immune effector cell-associated neurotoxicity syndrome (ICANs) | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, China